CLINICAL TRIAL: NCT06659406
Title: The Effect of Coenzyme Q10 Supplementation on Oxidative Stress, Inflammation and Hyperandrogenism in Women with Polycystic Ovary Syndrome
Brief Title: Effect of Coenzyme Q10 Administration on Polycystic Ovary Syndrome
Acronym: PCOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Collaborators: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, hira zahid, Assistant Professor, University of Faisalabad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Tuf/IRB/275/24
Record Dates: First submitted 2024-10-14; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CoQ-10 supplementation (Experimental): The experimental arm will consist of fertile females diagnosed with polycystic ovary syndrome aged between 18 to 50 years. Patients with diabetes mellitus, thyroid dysfunction, cardiovascular diseases, impairment of hepatic and renal function, autoimmune and Inflammatory disorders will be excluded.
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Coenzyme Q10 will be given once daily, 200mg for the period of 3 months
  Other Names: ubiquinone

SUMMARY:
The goal of this clinical trial is to determine the effects of coenzyme Q10 supplementation on oxidative stress, inflammation and hyperandrogenism in women with polycystic ovary syndrome. The main questions it aims to answer are:

Does Coenzyme Q10 alter oxidative stress, inflammation and hyperandrogenism in women with Polycystic ovary syndrome.

Participants will take Coenzyme Q10 200mg, once daily for a period of 3 months. The participants will be reassessed after 12 weeks by measuring Malondialdehyde MDA, C-reactive protein CRP, Sex hormone binding globulin SHBG.

ELIGIBILITY:
Inclusion Criteria:

* Married Patients that presented with anovulatory infertility due to PCOS.
* Unmarried Patients that presented with symptoms due to PCOS
* All patients should fulfill Rotterdam criteria for PCOS

Exclusion Criteria:

* Male factor infertility ( oligospermia or aspermia)
* Tubal factor infertility (abnormal hysterosalpingography)
* Diabetes mellitus, thyroid dysfunction, cardiovascular diseases, impairment of hepatic and renal function
* Autoimmune and Inflammatory disorders
* Abnormal serum prolactin level
* Smokers
* Alcoholic beverage use
* Use of anti diabetic, anti-obesity drugs, insulin or vitamin and mineral supplements

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological females would be accepted because this condition effects ovaries that are present in biological females only
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
effect of coenzyme q10 administration on polycystic ovary syndrome | from enrollment to the end of treatment at 12 weeks
  Improvement in levels of oxidative stress , inflammatory and hyperandrogenism biomarkers in women with Polycystic ovary syndrome
The effect of coenzyme Q10 supplementation on oxidative stress, inflammation and hyperandrogenism in women with polycystic ovary syndrome | from enrollment to the end of treatment at 12 weeks
  Oxidative stress in PCOS is leads to imbalance in antioxidant and oxidant levels in the body, along with production of reactive oxygen species. Insulin resistance has a key role in the PCOS pathogenesis by promoting oxidative stress and promoting acute and chronic Inflammation. Studies have shown that inflammatory markers are raised in PCOS along with decreased levels of anti-inflammatory biomarkers. Coenzyme Q10 is a natural vitamin, acts as an antioxidant, have shown an constructive impact on inflammatory and endothelial dysfunction biomarkers and also effects androgen levels. Effect of Coenzyme Q10 supplementation on oxidative stress, inflammation and hyperandrogenism will be accessed by biomarkers Malondialdehyde MDA, C-reactive protein CRP and Sex hormone binding globulin SHBG. Ideally levels of MDA, CRP would decrease and SHBG levels would increase after Coenzyme Q10 supplementation. This study would measure these three biomarkers before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Akram, MBBS, FCPS, Study Director — University of Faisalabad
Locations (1):
- Madinah Teaching Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
patients data will not be shared because it is highly confidential document

REFERENCES:
- [Background] Hu X, Wang W, Su X, Peng H, Tan Z, Li Y, Huang Y. Comparison of nutritional supplements in improving glycolipid metabolism and endocrine function in polycystic ovary syndrome: a systematic review and network meta-analysis. PeerJ. 2023 Nov 13;11:e16410. doi: 10.7717/peerj.16410. eCollection 2023. PMID 38025704
- See also: Efficacy of coenzyme Q10 supplementation on glucose metabolism, lipid profiles, and biomarkers of inflammation in women with polycystic ovary syndrome — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7668517/